CLINICAL TRIAL: NCT03128021
Title: Neural Mechanisms of Monoaminergic Engagement in Late-life Depression Treatment Response (NEMO)
Acronym: NEMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Howard Aizenstein (Other)
Collaborators: Weill Cornell Institute of Geriatric Psychiatry (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Howard Aizenstein, Charles F. Reynolds III and Ellen G. Detlefsen Endowed Chair in Geriatric Psychiatry and Associate Professor of Bioengineering and Clinical and Translational Science, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19120137; R01MH076079 (NIH)
Record Dates: First submitted 2017-04-04; First posted 2017-04-25 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression; fMRI; Escitalopram; Lexapro; Randomized Clinical Trial; Levomilnacipran; Fetzima
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Levomilnacipran

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to take either escitalopram or levomilnacipran throughout the 12-week trial.
  The following information applies to the original study design. Enrollment according to this design was complete as of April 2018: During Phase I, participants will be randomly assigned to take escitalopram or placebo daily for 6 weeks. After 6 weeks, participants who are randomly assigned to placebo will be given the option to have an open-label of escitalopram for Phase II. Those who did not respond to escitalopram in Phase I will be referred for alternate treatment. All participants, regardless of outcome will be asked to return for follow-up procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Although this is a double-blinded study, one staff member will be unblinded regarding study randomization. Should the need ever arise, the blind can be instantly broken for the participant's safety and well-being.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Escitalopram Pill (Active Comparator): Participants in this arm will receive an initial dose of 5 mg. Further titrations will be decided based on clinical response and tolerability (maximum dose of 20 mg). The medication will be taken by mouth in pill form, once daily.
  Interventions: Drug: Escitalopram Pill
- Placebo (Placebo Comparator): Participants will be given a sugar pill (placebo) to be taken by mouth once daily for the 6 week duration of Phase I. As this arm is also double-blinded, participants will receive an initial dose of 5 mg and further titrations (maximum dose of 20 mg) will be decided based on clinical response and tolerability.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima.
  Interventions: Other: Placebo
- Escitalopram Pill (Phase II) (Other): Participants who were in the placebo arm for Phase I who do not show signs of response to treatment by week 6 (defined as either a MADRS score of greater than 12 or less than a 30% reduction in MADRS score to be deemed a non-responder) will be given the option to have an open-label trial of escitalopram in Phase II.
  Participants in this arm will receive an initial dose of 5 mg. Further titrations throughout the 6 week duration of Phase 2 (maximum dose of 20 mg) will be decided based on clinical response and tolerability. The medication will be taken by mouth in pill form, once daily.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima and the assignment does not change throughout the study.
  Interventions: Drug: Escitalopram Pill
- Levomilnacipran Pill (Active Comparator): Participants will receive an initial dose of 20 mg blinded levomilnacipran. At day 7, the doses will be titrated to 40 mg of levomilnacipran. Further titrations (maximum dose of 120 mg of levomilnacipran) will be decided based on clinical response and tolerability. The medication will be taken by mouth in pill form, once daily.
  Interventions: Drug: Levomilnacipran Pill

INTERVENTIONS:
Drug: Escitalopram Pill — Double-blinded, randomly assigned
  Other Names: Lexapro
  Arms: Escitalopram Pill; Escitalopram Pill (Phase II)
Other: Placebo — Double-blinded, randomly assigned
  Arms: Placebo
Drug: Levomilnacipran Pill — Double-blinded, randomly assigned
  Other Names: Fetzima
  Arms: Levomilnacipran Pill

SUMMARY:
The Department of Psychiatry at the University of Pittsburgh is conducting a research study to learn about the changes that occur in the brain when individuals suffer from and then are treated for depression. The NEMO study has two main purposes. The first is to provide medication treatment to individuals ages 60 and older who are currently depressed.

The second part of the study involves completing a series of 4 MRIs, which assess changes in brain function over the course of treatment. This research may help investigators to develop faster and more effective treatment plans in the future, as brain responses that are detected early in treatment may predict how well an individual will respond to antidepressant medication.

DETAILED DESCRIPTION:
In this competing renewal (Year 11) of the investigators' R01 which has used functional magnetic resonance imaging (fMRI) to study late-life depression (LLD) pharmacotherapy (R01MH076079), the primary aim of this study is to characterize functional connectivity changes associated with initial medication exposure (12-hour challenge). Preliminary data suggests that these initial fMRI changes reflect monoaminergic engagement, regardless of monoaminergic class, and predict later treatment response. This study will test a neural systems level model that response in LLD is mediated by acute pharmacologically-induced changes in cognitive and affective large scale network.

Depression in older adults is frequently disabling and is often resistant to first-line treatments, requiring more prolonged treatment trials than in younger adults, mainly due to its heterogeneous pathophysiology (e.g. vascular and degenerative brain changes). Currently, there is little neurobiological data to guide changing or augmenting antidepressant medications. Thus, there has been a heightened focus on tailoring treatment to optimize outcome as described in the 2015 National Institute of Mental Health (NIMH) draft strategic plan (strategy 3.2). While antidepressant clinical response may take up to 8 weeks, recent studies suggest that physiologic changes, as measured with pharmacologic fMRI (phMRI) are seen within 12 hours of starting a new monoaminergic antidepressant (1).

For this proposal, investigators focus on three major Cognitive and Affective Networks (CAN): the Default Mode Network (DMN), the Salience Network (SN) and the Executive Control Network (ECN). The proposed model suggests that monoaminergic engagement leads to core CAN changes, changes that subsequently are related to overall clinical response as well as response in specific symptom clusters such as negative bias, somatizations/anxiety and cognitive control. The same networks that are functionally connected while individuals are at rest, are also selectively engaged during tasks. Investigators' prior work shows that pharmacotherapy - regardless of type of antidepressant used - engages these specific networks at rest and during standard cognitive and affective tasks. Given the role of cerebrovascular disease in LLD treatment response, the moderating role of vascular burden on the proposed association between CAN engagement and treatment response will also be explored.

The University of Pittsburgh will recruit 100 older adults with LLD that will be randomized to receive treatment with either a very specific serotonin reuptake inhibitor (escitalopram) or a norepinephrine reuptake inhibitor (levomilnacipran). A pair of fMRI scans one day apart will be used to measure functional connectivity (FC) associated with medication titration. Investigators will use a very early (12 hours after initiation of treatment) biomarker of treatment response, which, when validated, would decrease substantially the waiting time between medication changes. Additionally, this study will further increase knowledge of the acute neural system changes associated with monoaminergic antidepressants; this knowledge of mechanism is essential for both guiding LLD treatment research, and serving as an engagement target in LLD treatment research.

Note: The original study design involved randomization to escitalopram or placebo (instead of escitalopram and levomilnacipran). Therefore a subset of participants will complete the study according to this design.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years old
* Current Major Depressive Episode or Current Depressive Disorder Not Otherwise Specified or Dysthymic Disorder
* Montgomery-Asberg Depression Rating Scale (MADRS) greater than or equal to 12
* Modified Mini-Mental State (3MS) score greater than or equal to 84
* MoCA-BLIND greater than or equal to 13

Exclusion Criteria:

* History of Mania or Psychosis
* Current suicidal ideation that cannot be safely managed within the confines of a clinical trial
* Alcohol or Substance Abuse (current or past 3 months) endorsed via phone screening interview or diagnosed by Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID)
* Dementia of any etiology endorsed via phone screening interview or diagnosed by SCID
* Medical conditions with known significant effects on mood (e.g., stroke, current hypothyroid state) as well as unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cardiovascular risk factors that are not under medical management Unwilling or clinically determined to be unable to taper from high doses of benzodiazepines (equivalent to > 2 mg lorazepam/day) or other anti-depressant/anti-anxiety medications at time of screening. However, for participants who are prescribed low dose psychotropics for pain, sleep disturbances, and/or medical conditions (e.g. amitriptyline for peripheral neuropathy, low dose trazodone as a sleep aid), these will be allowed in most circumstances. We will include participants on certain dosages of the most commonly prescribed antidepressants (for medical reasons) as follows: amitriptyline up to 50 mg/d, doxepin up to 50 mg/d, trazodone up to 100 mg/d, and imipramine up to 50 mg/d. Participants will also be able to continue taking buspirone, an antianxiety medication. As per the examples above, the PI will decide if the participants are eligible for the study and if they may continue the current medication. Justification regarding all decisions will be documented in the research record.
* Inability to complete required assessments including brain MRI and blood draw
* Hearing/vision impairment precluding neuropsychological testing
* Difficulty conversing in English
* Clinical contraindication to use of escitalopram or levomilnacipran or history of treatment resistance to escitalopram or levomilnacipran
* Unable or unwilling to provide a secondary/emergency contact person
* History of stroke with residual symptoms, current epilepsy, or current post-concussive symptoms
* Clinically relevant hyponatremia (below 130 mEq/L)
* Significant renal impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard J Aizenstein, MD, Ph.D., Principal Investigator — Charles F. Reynolds III and Ellen G. Detlefsen Endowed Chair in Geriatric Psychiatry and Associate Professor of Bioengineering and Clinical and Translational Science; Carmen Andreescu, MD, Principal Investigator — Assistant Professor of Psychiatry
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared through the NIMH Data Archive.
Time Frame: Data collected to date is submitted twice annually (January and July) and is shared within 4 months of submission.
Access Criteria: NIH will provide access to scientific investigators for research purposes.
URL: https://ndar.nih.gov/edit_collection.html?id=2583

REFERENCES:
- [Background] Andreescu C, Reynolds CF 3rd. Late-life depression: evidence-based treatment and promising new directions for research and clinical practice. Psychiatr Clin North Am. 2011 Jun;34(2):335-55, vii-iii. doi: 10.1016/j.psc.2011.02.005. PMID 21536162
- [Background] Delis DC, Kaplan, E., Kramer, J.H. Delis Kaplan Executive Funciton System Examiner's Manual. The Psychological Corporation; 2001.
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Tomaszewski Farias S, Mungas D, Harvey DJ, Simmons A, Reed BR, Decarli C. The measurement of everyday cognition: development and validation of a short form of the Everyday Cognition scales. Alzheimers Dement. 2011 Nov;7(6):593-601. doi: 10.1016/j.jalz.2011.02.007. PMID 22055976
- [Background] Isella V, Villa L, Russo A, Regazzoni R, Ferrarese C, Appollonio IM. Discriminative and predictive power of an informant report in mild cognitive impairment. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):166-71. doi: 10.1136/jnnp.2005.069765. PMID 16421116

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will be given a sugar pill (placebo) to be taken by mouth once daily for the 6 week duration of Phase I. As this arm is also double-blinded, participants will receive an initial dose of 5 mg and further titrations (maximum dose of 20 mg) will be decided based on clinical response and tolerability.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima.
  Placebo: Double-blinded, randomly assigned
- Escitalopram Pill (Phase II): Participants who were in the placebo arm for Phase I who do not show signs of response to treatment by week 6 (defined as either a MADRS score of greater than 12 or less than a 30% reduction in MADRS score to be deemed a non-responder) will be given the option to have an open-label trial of escitalopram in Phase II.
  Participants in this arm will receive an initial dose of 5 mg. Further titrations throughout the 6 week duration of Phase 2 (maximum dose of 20 mg) will be decided based on clinical response and tolerability. The medication will be taken by mouth in pill form, once daily.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima and the assignment does not change throughout the study.
  Escitalopram Pill: Double-blinded, randomly assigned
Period: Overall Study
Arm/Group | Escitalopram Pill | Placebo | Escitalopram Pill (Phase II) | Levomilnacipran Pill
Started | 25 | 4 | 6 | 22
Completed | 20 | 2 | 4 | 9
Not Completed | 5 | 2 | 2 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram Pill | Placebo | Escitalopram Pill (Phase II) | Levomilnacipran Pill | Total
Number analyzed (Participants) | 25 | 4 | 6 | 22 | 57
Age, Continuous [Mean (Standard Deviation); unit: age at randomzation] | 68.13 (6.29) | 63.74 (3.02) | 64.47 (2.17) | 68.43 (7.72) | 67.55 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 5 | 10 | 31
  Male | 12 | 1 | 1 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 24 | 4 | 6 | 22 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 3 | 11
  White | 22 | 2 | 3 | 18 | 45
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 4 | 6 | 22 | 57
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Montgomery Asberg Depression Rating Scale measures depression severity. Scores can range from 0 to 60, with higher scores indicating higher levels of depression severity. Population: 8 participants were eligible after screening measures, were randomized, but were then terminated from the study before "baseline" MADRS scores were recorded.
  units on a scale
    number analyzed (Participants) | 23 | 3 | 6 | 17 | 49
    (all) | 19.43 (6.68) | 25.33 (5.51) | 23.83 (5.19) | 21.94 (6.35) | 21.20 (6.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale Score
Description: Treatment response will be defined as either a MADRS score of less than 12 or 30% or greater reduction in MADRS score.
Time Frame: Change in Baseline MADRS score through Week 12
Measure: Number; unit: persons with positive treatment response
Arm/Group | Escitalopram Pill | Placebo | Escitalopram Pill (Phase II) | Levomilnacipran Pill
Number analyzed (Participants) | 20 | 2 | 4 | 9
persons with positive treatment response | 18 | 2 | 3 | 8

2. Primary Outcome: Change in Functional Connectivity
Description: The primary analysis will consist of linear mixed effects models with functional connectivity (for each region of interest) as the outcome measure and group (R [responder]/NR[non-responder], as defined by MADRS), time and their interaction.
  The results listed are the difference in Baseline to 12 hours after first dose of medication.
  The values derived by first preprocessing the raw data using SPM and using the AAL3 atlas to parcellate the images into anatomical brain regions. Then the mean residual time series for each region was calculated and the Pearson correlation between the time series of each region was calculated. Then the mean Pearson correlations between every other region with the region identified were calculated and these correlation values were then standardized to have a mean of 0 and a standard deviation of 1. Higher values indicate stronger and better connectivity.
Time Frame: Change in Functional Connectivity from Baseline to Day 1
Population: Total participants with available Baseline and Day 1 scans that could be analyzed.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Escitalopram Pill (R); Escitalopram Pill (NR): Participants in this arm will receive an initial dose of 5 mg. Further titrations will be decided based on clinical response and tolerability (maximum dose of 20 mg). The medication will be taken by mouth in pill form, once daily.
  Escitalopram Pill: Double-blinded, randomly assigned
- Placebo (R): Participants will be given a sugar pill (placebo) to be taken by mouth once daily for the 6 week duration of Phase I. As this arm is also double-blinded, participants will receive an initial dose of 5 mg and further titrations (maximum dose of 20 mg) will be decided based on clinical response and tolerability.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima.
  Placebo: Double-blinded, randomly assigned
- Escitalopram Pill (R) (Phase II); Escitalopram Pill (NR) (Phase II): Participants who were in the placebo arm for Phase I who do not show signs of response to treatment by week 6 (defined as either a MADRS score of greater than 12 or less than a 30% reduction in MADRS score to be deemed a non-responder) will be given the option to have an open-label trial of escitalopram in Phase II.
  Participants in this arm will receive an initial dose of 5 mg. Further titrations throughout the 6 week duration of Phase 2 (maximum dose of 20 mg) will be decided based on clinical response and tolerability. The medication will be taken by mouth in pill form, once daily.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima and the assignment does not change throughout the study.
  Escitalopram Pill: Double-blinded, randomly assigned
- Levomilnacipran Pill (R); Levomilnacipran Pill (NR): Participants will receive an initial dose of 20 mg blinded levomilnacipran. At day 7, the doses will be titrated to 40 mg of levomilnacipran. Further titrations (maximum dose of 120 mg of levomilnacipran) will be decided based on clinical response and tolerability. The medication will be taken by mouth in pill form, once daily.
  Levomilnacipran Pill: Double-blinded, randomly assigned
- Placebo (NR): Participants will be given a sugar pill (placebo) to be taken by mouth once daily for the 6 week duration of Phase I. As this arm is also double-blinded, participants will receive an initial dose of 5 mg and further titrations (maximum dose of 20 mg) will be decided based on clinical response and tolerability.
  Note: This arm no longer applies as of 5/16/18. Participants are now randomly assigned to Lexapro or Fetzima.
Arm/Group | Escitalopram Pill (R) | Placebo (R) | Escitalopram Pill (R) (Phase II) | Levomilnacipran Pill (R) | Escitalopram Pill (NR) | Placebo (NR) | Escitalopram Pill (NR) (Phase II) | Levomilnacipran Pill (NR)
Number analyzed (Participants) | 15 | 0 | 5 | 7 | 2 | 0 | 1 | 0
Z-score
  Left Middle Frontal Gyrus day 1 difference | 0.059122257 (0.970768475) |  | -0.337856865 (0.456280057) | -0.682262788 (0.394139675) | -0.005553818 (0.336358139) |  | -0.577911771 |
  Right Middle Frontal Gyrus day 1 difference | 0.090272305 (1.047858325) |  | 0.80863611 (0.591200619) | -0.064993511 (0.942271068) | 1.243841088 (0.160518864) |  | -1.315813839 |
  Left Anterior Insular day 1 difference | 0.007749148 (1.206679758) |  | -0.48413394 (1.3756677) | -0.224292239 (0.655920209) | -1.553051837 (0.638678017) |  | 0.976927111 |
  Right Anterior Insular day 1 difference | -0.227766723 (1.228475106) |  | -0.23236189 (0.616824453) | 0.147147958 (0.887236616) | 1.056817365 (1.504505678) |  | 0.820792593 |
  Left Amygdala day 1 difference | 0.259715101 (0.91863688) |  | -0.592134869 (1.3814767) | 0.147597427 (0.599482713) | -1.33405492 (0.601671616) |  | 1.9845321 |
  Right Amygdala day 1 difference | -0.443833224 (1.739580169) |  | -1.311685475 (1.328056717) | 0.548047987 (1.379828096) | -0.030660361 (0.159008845) |  | 0.964444893 |
  Left prefrontal Anterior Cingulate Cortex day 1 difference | 0.048557684 (1.079632973) |  | 0.735636432 (1.010043826) | -0.003163926 (0.783815631) | -0.216753695 (0.608987758) |  | -1.215843301 |
  Right prefrontal Anterior Cingulate Cortex day 1 difference | 0.206183452 (1.994469683) |  | 1.413900498 (1.543971432) | 0.131919092 (0.80516401) | 0.839416177 (2.093317463) |  | -1.637127786 |

3. Secondary Outcome: Response Styles Questionnaire- Rumination (RSQ-Rumination)
Description: The Response Styles Questionnaire- Rumination (RSQ-Rumination) examines propensity towards negative bias during thought. To be used as covariate in functional connectivity analysis.
  Range of scores: 22-88. Lower the better
Time Frame: Baseline, Week 1, and Week 12
Population: Participants who completed all 12 weeks of the study with RSQ scores.
Measure: Mean (Standard Deviation); unit: RSQ total score
Arm/Group | Escitalopram Pill (R) | Placebo (R) | Escitalopram Pill (R) (Phase II) | Levomilnacipran Pill (R) | Escitalopram Pill (NR) | Placebo (NR) | Escitalopram Pill (NR) (Phase II) | Levomilnacipran Pill (NR)
Number analyzed (Participants) | 15 | 2 | 3 | 8 | 2 | 0 | 1 | 1
RSQ total score
  Baseline | 45.1 (11.01) | 39.5 (3.54) | 60.7 (11.15) | 49.7 (8.73) | 67.5 (.071) |  | 49 | 50
  Week 01 | 39 (11.08) | 40.5 (2.12) | 52.3 (16.74) | 40.5 (7.23) | 61 (9.90) |  | 46 | 51
  Week 12 | 33.7 (10.39) | 28.5 (3.54) | 42.7 (8.96) | 40.4 (9.87) | 60 (1.41) |  | 30 | 67

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HARS)
Description: The Hamilton Anxiety Rating Scale (HARS) is a structured interview to assist in the reliable assessment of anxiety severity by standardizing the method of assessment and providing clear anchor points for the assignment of severity ratings. Examines level of anxiety and somatization. To be used as covariate in functional connectivity analysis.
  Range of scores: 0-56. Lower the better
Time Frame: Baseline, Week 1, and Week 12
Population: Participants who completed all 12 weeks of the study with HARS scores.
Measure: Mean (Standard Deviation); unit: HARS total score
Arm/Group | Escitalopram Pill (R) | Placebo (R) | Escitalopram Pill (R) (Phase II) | Levomilnacipran Pill (R) | Escitalopram Pill (NR) | Placebo (NR) | Escitalopram Pill (NR) (Phase II) | Levomilnacipran Pill (NR)
Number analyzed (Participants) | 16 | 2 | 3 | 8 | 2 | 0 | 1 | 1
HARS total score
  Baseline | 19.3 (6.66) | 22.5 (9.19) | 26.6 (3.05) | 21.5 (5.26) | 25.5 (2.12) |  | 24 | 23
  Week 01 | 12.3 (6.40) | 19.5 (7.78) | 18.3 (7.64) | 16.4 (4.53) | 21.5 (3.54) |  | 17 | 24
  Week 12 | 7.5 (5.44) | 7 (5.66) | 19.7 (1.53) | 10.6 (8.33) | 18.5 (4.95) |  | 20 | 32

5. Secondary Outcome: Neuropsychological Evaluations
Description: The neuropsychological testing battery, developed by Co-I Meryl Butters, Ph.D., includes components of the Delis-Kaplan Executive Function Scale (D-KEFS), and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
  "dkefs_trail4_scaled_1" is a scaled score for Condition 4 (Number-Letter Switching) of the D-KEFS Trail Making Test, which measures cognitive flexibility and executive functioning. Range 1-19. Higher the better
  " dkefs_colorword3_scaled_1" is a score from D-KEFS Color-Word Interference. The individual is asked to inhibit an automatic reading response to name the ink color of words that spell out conflicting color names. Range 1-19. Higher the better
  "rbans_total_index_1" is the total index score from the RBANS, designed to assess various cognitive domains. The total index score is a composite score that provides an overall measure of cognitive functioning by combining the results from all the RBANS subtests. Range 40-155. Higher the better
Time Frame: Baseline and Week 12
Population: Participants who had complete neuropsychological testing at both Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram Pill | Levomilnacipran Pill | Placebo | Escitalopram Pill (Phase II)
Number analyzed (Participants) | 10 | 1 | 2 | 5
score on a scale
  dkefs_trail4_scaled_1_Baseline | 11 (3.71) | 11 | 8 (5.66) | 10.6 (3.21)
  dkefs_trail4_scaled_1_Week12 | 10.8 (3.65) | 11 | 9 (4.24) | 12.25 (1.26)
  dkefs_colorword3_scaled_1_Baseline | 11 (3.26) | 9 | 9 (0) | 11 (2.00)
  dkefs_colorword3_scaled_1_Week12 | 11.6 (2.50) | 9 | 10.5 (0.71) | 10.6 (3.58)
  rbans_total_index_1_Baseline | 97.4 (9.21) | 110 | 94 (1.41) | 103.2 (17.92)
  rbans_total_index_1_Week12 | 102.9 (12.04) | 107 | 102.5 (2.12) | 102.6 (20.41)

6. Secondary Outcome: Antidepressant Treatment History Questionnaire (ATHF)
Description: Investigators will examine prior treatment history and how this may affect treatment response in this study. Number of participants analyzed are those who have previously had a trial of at least one antidepressant.
Time Frame: Baseline
Population: The Outcome are those who were considered "responders" for this study. No participants in the Placebo group had previously taken an antidepressant.
Measure: Count of Participants; unit: Participants
Arm/Group | Escitalopram Pill | Placebo | Escitalopram Pill (Phase II) | Levomilnacipran Pill
Number analyzed (Participants) | 9 | 0 | 2 | 3
Participants | 7 | 0 | 1 | 2

7. Secondary Outcome: Medication Plasma Levels
Description: Investigators will assess how blood levels of escitalopram and levomilnacipran may affect treatment response.
  The data was not collected because the Co-Investigator responsible for the analyses left academia and the University of Pittsburgh. No data will ever be produced and there will be no results to report.
Time Frame: Weeks 1-12
Population: Analyses will not be performed at any time in the future.
Arm/Group | Escitalopram Pill | Levomilnacipran Pill | Placebo | Escitalopram Pill (Phase II)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Age of Onset
Description: Investigators will assess how early vs. late onset depression (e.g., onset before/after age 60) may affect treatment response.
Time Frame: Baseline
Population: Age of onset for current depressive episode and how it relates treatment outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Escitalopram Pill (R) | Placebo (R) | Escitalopram Pill (R) (Phase II) | Levomilnacipran Pill (R) | Escitalopram Pill (NR) | Placebo (NR) | Escitalopram Pill (NR) (Phase II) | Levomilnacipran Pill (NR)
Number analyzed (Participants) | 16 | 2 | 3 | 6 | 2 | 0 | 0 | 1
Participants
  Number of participants age of onset before age 60 | 6 | 2 | 2 | 2 | 2 | 0 | 0 | 1
  Number of participants age of onset at or after age 60 | 10 | 0 | 1 | 4 | 0 | 0 | 0 | 0

9. Secondary Outcome: Duration of Illness
Description: Investigators will assess how length of current episode affect treatment response.
Time Frame: Duration of illness at Baseline
Population: Number of participants analyzed if information was available during interviews
Measure: Count of Participants; unit: Participants
Arm/Group | Escitalopram Pill (R) | Placebo (R) | Escitalopram Pill (R) (Phase II) | Levomilnacipran Pill (R) | Escitalopram Pill (NR) | Placebo (NR) | Escitalopram Pill (NR) (Phase II) | Levomilnacipran Pill (NR)
Number analyzed (Participants) | 16 | 2 | 3 | 6 | 2 | 0 | 0 | 1
Participants
  Duration of one year or less | 6 | 0 | 1 | 3 | 0 | 0 | 0 | 1
  Duration of more than one year to 10 years | 5 | 0 | 0 | 2 | 2 | 0 | 0 | 0
  Duration of more than 10 years | 5 | 2 | 2 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Escitalopram Pill | Levomilnacipran Pill | Placebo | Escitalopram Pill (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 13/25 | 6/22 | 0/4 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram Pill (N=25) | Levomilnacipran Pill (N=22) | Placebo (N=4) | Escitalopram Pill (Phase II) (N=6)
anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
drowsiness or yawning (General disorders) | 10 (16) | 2 (3) | 0 (0) | 3 (3)
dry mouth (General disorders) | 6 (6) | 3 (3) | 0 (0) | 2 (2)
extrapyramidal symptoms (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
headache (General disorders) | 7 (7) | 5 (5) | 0 (0) | 2 (2)
heartburn (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
increased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
increased body temperature/sweating (General disorders) | 5 (6) | 2 (3) | 0 (0) | 1 (1)
increased irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
increased sleep (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
insomnia or trouble sleeping (General disorders) | 8 (8) | 4 (4) | 0 (0) | 2 (2)
lightheadedness (General disorders) | 5 (7) | 5 (6) | 0 (0) | 0 (0)
nausea or vomiting (General disorders) | 6 (7) | 5 (5) | 0 (0) | 2 (2)
palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
rash/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
uninary problems (Renal and urinary disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0)
vertigo (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
weight gain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03128021/Prot_SAP_000.pdf